CLINICAL TRIAL: NCT05429671
Title: Drug Elution Profile and Minimum Inhibitory Concentration of Antibiotic-loaded Cement After Primary Total Knee Arthroplasty
Brief Title: Antibiotic Loaded Cement After TKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAUS21D.1213
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Total Knee Arthoplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee; Tobramycin; Gentamicins

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group A (Control-negative group) (Active Comparator): include participants undergoing total knee arthroplasty with Stryker Surgical Simplex P cement containing no antibiotic
  Interventions: Procedure: total knee arthroplasty
- Group B (tobramycin group) (Active Comparator): includes participants undergoing total knee arthroplasty with Stryker Surgical Simplex P cement with tobramycin antibiotic.
  Interventions: Procedure: total knee arthroplasty; Drug: Tobramycin
- Group C (gentamicin group) (Active Comparator): Include participants undergoing total knee arthroplasty with Huraeus Palacos R+G cement containing gentamicin antibiotic.
  Interventions: Procedure: total knee arthroplasty; Drug: Gentamicin
- Group D (Control-positive group) (Active Comparator): Include participants undergoing the first of a two-stage exchange arthroplasty for confirmed infection, using an antibiotic-loaded cement spacer. These patients will have a spacer implant made of vancomycin and tobramycin antibiotics using Huraeus Palacos non-antibiotic loaded cement
  Interventions: Procedure: total knee arthroplasty; Device: Antibiotic cement spacer

INTERVENTIONS:
Procedure: total knee arthroplasty — Participants will have total knee arthroplasty
Drug: Tobramycin — Total knee arthroplasty using Stryker Surgical Simplex P with tobramycin
  Arms: Group B (tobramycin group)
Drug: Gentamicin — Total knee arthroplasty using Huraeus Palacos R+G cement containing gentamicin
  Arms: Group C (gentamicin group)
Device: Antibiotic cement spacer — participants getting an antibiotic-loaded cement spacer during surgery comprised of vancomycin and tobramycin.
  Arms: Group D (Control-positive group)

SUMMARY:
This study will provide us with clear information about the postoperative concentration of antibiotic reached in synovial fluid, thereby helping surgeons to determine if concentration could potentially prevent the growth and regrowth of common infecting microorganisms (based on their MIC and MBEC). There is a need to define the actual benefit of antibiotic-loaded bone cement, because the addition of antibiotic can reduce its mechanical strength. Moreover, if sub-therapeutic antibiotic levels are achieved, this could facilitate the emergence of resistant bacterial strains. Amidst the transition towards value-based care, our research will enable surgeons to decide whether antibiotic-loaded cement is truly cost-effective in the prevention of PJI.

ELIGIBILITY:
Inclusion Criteria:

* All participants undergoing cemented primary total knee arthroplasty (TKA) who are 18 years or older.

Exclusion Criteria:

* Withdrawal of informed consent,
* allergy to any of the study medications or to bone cement,
* use of antibiotics within 4 weeks before collecting the samples (not including perioperative antimicrobial prophylaxis),
* high risk of infection,
* history of peri-articular injections for multimodal pain management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Antibiotic concentration | 24 hours
  To determine antibiotic levels, synovial fluid (joint fluid) would be taken after surgery to measure the concentration of antibiotic in the joint fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States